CLINICAL TRIAL: NCT05377710
Title: Multicentre, Interventional, Longitudinal, Open-label Study Conducted in France Evaluating the Clinical Performance and Safety of Glycobone® as a Bone Filler in a Lateral Sinus Lift Setting
Brief Title: Evaluation of the Safety and Performance of Glycobone in Sinus Lift
Acronym: SL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SILTISS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A02457-32
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Sinus Elevation; Bone Substitute

STUDY DESIGN:
Intervention Model Description: human
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glycobone (Experimental): Patients will be implanted at T0 with Glycobone
  Interventions: Procedure: sinus lift with lateral approach

INTERVENTIONS:
Procedure: sinus lift with lateral approach — Maxillary sinus floor augmentation or sinus lift is a surgical procedure, which provides a solution to the problem of sinus bone loss (too thin), and thus increases the thickness of the bone for immediate or subsequent implant placement in the premolars and molars (4). It consists of the elevation of the sinus mucosa that lines the maxillary sinus. The space thus freed will be filled with a bone filling material
  Other Names: sinus elevation

SUMMARY:
Multicentre, interventional, longitudinal, open-label study conducted in France, evaluating the clinical performance and safety of Glycobone® as a bone filling material in the context of a lateral approach sinus lift on 40 patients with dental implant placement. Implant placement took place 6 months after bone filling.

DETAILED DESCRIPTION:
A multicentre, interventional, longitudinal, open-label, prospective, pilot exploratory study of first-in-man administration in France, evaluating the clinical performance, safety and bone filling properties of Glycobone® during a lateral sinus lift procedure with deferred implant placement.

The study will follow a panel of 40 patients for 9 months in three consecutive stages:

Stage 1: Inclusion of a group of up to 5 patients Stage 2: If safety validation in stage 1 is confirmed: Inclusion of a group of 15 additional patients (maximum) Step 3: If safety validation in step 2 is confirmed: Inclusion of a group of 20 additional patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patient, male or female, aged 18-84 years at the time of signing the consent form

  2. Patient who has been informed and has signed consent prior to any procedure related to the investigation 3. Patient requiring a dental implant procedure:
* Implant project associated with at least one lateral approach sinus lift due to sub-sinus bone height < 5 mm, without full bridge
* Associated with a bone filling
* With implant placement deferred to approximately 6 months within the limit of a maximum of 3 implants in the framework of the investigation 4. Availability of a cone beam with radiological guide less than 3 months old 5. Patient covered by a health insurance plan.

Exclusion Criteria:

1. 3 months or less old tooth extraction (≤ 3 months)
2. Sinus lift project requiring placement of all contralateral implants at the same time (i.e. 2 sinus lift projects associated with a full bridge)
3. Contralateral sinus lift of the site to be included performed within 3 months prior to inclusion
4. 4. Patient's general condition does not allow the investigator to perform the investigative procedures
5. Pregnant or breastfeeding patient at the time of the sinus lift and filling procedure (D0)
6. Patient with a concomitant ENT infection that may interfere with the investigative procedures
7. Patient with an uncontrolled chronic condition that may interfere with investigative procedures
8. Patient on VKA with INR >4, biphosphonates, denosumab or having been treated with radiotherapy in the study area
9. Patient unable to receive any type of analgesic during the investigation
10. Patient allergic to any of the components of Glycobone®.
11. Patient participating or having participated in another drug or medical device clinical trial within 30 days prior to inclusion in this study
12. Patient considered by the investigator to be non-compliant with study procedures
13. Patient deprived of liberty by court or administrative order or under legal protection (e.g. guardianship)

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-16 (Estimated); Primary Completion 2022-05-16 (Estimated); Study Completion 2022-05-16 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the success rate of the implantation at 6 months | 6 months after implantation
  The primary endpoint of the investigation is the success rate at M6 defined as the number of successfully placed implants (with sufficient bone formation judged by the implantologist and an implant judged to be stable) compared to the total number of implants planned to be placed at the beginning of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean PAUFIQUE, Study Director — SILTISS; Sylvain CATROS, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No
It is a private study belonging to SILTISS; the data will not be transmitted to other scientists but will remain within SILTISS to be valorised